CLINICAL TRIAL: NCT06779253
Title: An Open-label, Fixed-Sequence Study to Investigate The Effect of Multiple Oral Doses of Pimicotinib on The Pharmacokinetics of Metformin, Fexofenadine and Rosuvastatin In Healthy Subjects
Brief Title: A Study to Investigate The Effect of Pimicotinib on The Pharmacokinetics of Metformin, Fexofenadine and Rosuvastatin In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ABSK021-110
Record Dates: First submitted 2025-01-09; First posted 2025-01-16 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: Fexofenadine and rosuvastatin will be administered together as a cocktail, and metformin will be given via staggered dosing from the cocktail drugs administration. All subjects will receive the following study interventions:Day 1: metformin； Day 3: cocktail；Day 8 to 13: pimicotinib once daily (QD)；Day 14: metformin + pimicotinib；Day 15: pimicotinib，Day 16: cocktail + pimicotinib，Day 17 to 20: pimicotinib QD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pimicotinib with Metformin, Fexofenadine and Rosuvastatin (Other): Multiple oral doses of pimicotinib (50 mg QD) on the pharmacokinetics of fexofenadine (P-gp sensitive substrate), rosuvastatin (BCRP sensitive substrate) and metformin (MATE1 sensitive substrate). Fexofenadine and rosuvastatin will be administered together as a cocktail, and metformin will be given via staggered dosing from the cocktail drugs administration.All subjects will receive the following study interventions:Day 1: metformin, Day 3: cocktail, Day 8 to 13: pimicotinib once daily (QD), Day 14: metformin + pimicotinib, Day 15: pimicotinib, Day 16: cocktail + pimicotinib, Day 17 to 20: pimicotinib QD
  Interventions: Drug: pimicotinib capsules

INTERVENTIONS:
Drug: pimicotinib capsules — the effect of multiple oral doses of pimicotinib (50 mg QD) on the pharmacokinetics of fexofenadine (P-gp sensitive substrate), rosuvastatin (BCRP sensitive substrate) and metformin (MATE1 sensitive substrate). Fexofenadine and rosuvastatin will be administered together as a cocktail, and metformin will be given via staggered dosing from the cocktail drugs administration

SUMMARY:
This is a an open-label, fixed-sequence DDI study conducted in Chinese healthy subjects to investigate the effect of multiple oral doses of pimicotinib on the pharmacokinetics of fexofenadine , rosuvastatin and metformin . Fexofenadine and rosuvastatin will be administered together as a cocktail, and metformin will be given via staggered dosing from the cocktail drugs administration.

Approximately 38 healthy subjects will be enrolled to achieve 28 evaluable healthy subjects complete the study.

Blood samples will be collected for PK analysis .

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged 18 to 50 years (inclusive) at screening and at least 25% of each sex should be included.
2. Weight ≥ 50.0 kg (male) or ≥ 45.0 kg (female), with a body mass index (BMI) between 18.0 and 28.0 (inclusive), BMI = weight (kg)/height (m)2;
3. Normal or abnormal but not clinically significant results in physical examination, clinical laboratory tests and other relevant examinations as assessed by the investigator at Screening;
4. Male or female subjects of childbearing potential must agree to use effective methods of contraception during the study and within 6 months after the last dose of investigational product, and male subjects should not donate sperm during such period; female subjects should not donate ovum during such period and should not be pregnant or lactating. Pregnancy period is defined as the period from the date of conception until termination of pregnancy, and will be determined by laboratory test of human chorionic gonadotropin (hCG) during medical examination and baseline prior to initiation of the study;
5. Willing to participate in this study, understand the study procedures and sign the informed consent form prior to screening; willing to comply with the study procedures.

   -

Exclusion Criteria:

1. Past or current medical history of chronic or severe conditions in cardiovascular, respiratory, blood, liver, kidney, gastrointestinal, endocrine or nervous systems;
2. Known or persistent mental disorders that may preclude the participant from participation in the study, as determined by the investigator;
3. Past history of gastric or intestinal surgery, or other operations (except for appendectomy) affecting the drug absorption;
4. Dysphagia or inability to take the investigational product orally;
5. Intolerant to venipuncture, difficult to collect blood samples, or fear of needle sickness and blood;
6. Known allergy to two or more kinds of foods and drugs; or allergic to fexofenadine, rosuvastatin, metformin or pimicotinib or its excipients (lactose monohydrate, microcrystalline cellulose, colloidal silicon dioxide, croscarmellose sodium, magnesium stearate, gelatin, titanium dioxide); and prone to allergic reactions such as rash and urticaria;
7. History of bacterial, fungal, parasitic, viral (excluding nasopharyngitis), mycobacterial infection, and COVID-19 infection within 30 days prior to screening; or abnormal chest X-ray finding, assessed as clinically significant (by the investigator);
8. Symptoms of fatigue and pyrexia within 2 weeks prior to screening;
9. Abnormal laboratory tests;
10. Positive result for either of the following tests: serum Hepatitis B Surface Antigen (HBsAg), Hepatitis C Virus (HCV) antibody, Human Immunodeficiency Virus (HIV) antibody, and treponema pallidum antibody;
11. Participated in any clinical studies of drugs as a study participant and received the study drug within 3 months prior to screening;
12. Previously participated in any other study related to pimicotinib and received pimicotinib;
13. Used strong inhibitors or inducers of CYP3A4(including grapefruit juice, grapefruit hybrids, punica granatum, carambola, citrus maxima, and Seville oranges) and transporter P-gp/BCRP/MATE1/OATP1B1/OATP1B3/MATE2-K/OCT2 inhibitors within 14 days prior to screening and at Screening or intending to use during the study;
14. Have special dietary requirements or cannot accept to take a unified diet; specific dietary requirements: the subjects can only eat the food provided by the study site during hospitalization;
15. Consumption of more than 14 units of alcohol per week (1 unit of alcohol = about 360 mL of beer or 45 mL of spirits containing 40% alcohol or 150 mL of wine) within 3 months prior to signing the informed consent form, or a positive result for alcohol breath test on the day pre-dose (breath alcohol content > 0.0 mg/100 mL), or unable to abstain from alcohol during the study;
16. Consumption of more than 5 cigarettes per day within 3 months prior to signing the informed consent form, or unable to abstain from tobacco products during the study;
17. Previous chronic consumption of excessive amount of tea, coffee, or caffeinated beverages (excessive intake is defined as taking more than 6 units of caffeine per day, 1 unit of caffeine equivalent to 177 mL of coffee, 355 mL of tea, 355 mL of cola, or 85 g of chocolate) or unable to abstain from caffeinated beverages during the study;
18. Known history of drug abuse or positive for drug abuse screening test (morphine, methamphetamine, ketamine, methylene dioxyamphetamine, and tetrahydrocannabinol acid);
19. Used over the counter or prescription drugs, including herbal medicine, health products, vitamins, and dietary supplements, within 14 days prior to screening, or plan to use such drugs during the study;
20. Donated or lost > 400 mL of blood within 3 months prior to screening; received blood transfusions or used blood products within 2 months prior to screening;
21. Received vaccine (including COVID-19 vaccine) within 2 months prior to screening, or plan to get vaccinated during the study;
22. Abnormalities in vital signs (only one retest was allowed), including: ear temperature > 37.2 ℃; pulse rate > 100 beats/min or < 55 beats/min; systolic blood pressure ≥ 140 mmHg or < 90 mmHg, diastolic blood pressure ≥ 90 mmHg or <60 mmHg;
23. Heart rate-corrected QT interval prolongation, QTcF > 450 ms for males (> 470 ms for females) (Note: QTc interval corrected using the Fridericia formula), or family history of long QT syndrome, or other clinically significant ECG abnormalities at Screening;
24. Subjects involved in the design or conduct of this study and their immediate family members ;
25. Subjects who, in the opinion of the investigator, are not suitable for enrollment or may not be able to complete the study for other reasons.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Cmax | pre-dose, post-dose 0.5 hour, 1 hour, 1.5hours,2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours
  Peak concentration, the maximum observed plasma concentration of metformin, fexofenadine and rosuvastatin
AUClast | pre-dose, post-dose 0.5 hour, 1 hour, 1.5hours,2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours
  Area under the plasma concentration-time curve from time 0 to the time of last measurable concentration
AUC0-∞ | pre-dose, post-dose 0.5 hour, 1 hour, 1.5hours,2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours
  Area under the plasma concentration-time curve from time 0 to infinity

SECONDARY OUTCOMES:
AE | through study completion, an average of 50 days
  Safety profile of pimicotinib in combination with metformin, fexofenadine and rosuvastatin including but not limited to Adverse events (AEs),

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Doctor, Principal Investigator — The First Affiliated Hospital Shandong First Medical University (Shandong Provincial Qianfoshan Hospital)
Locations (1):
- The First Affiliated Hospital Shandong First Medical University (Shandong Provincial Qianfoshan Hospital), Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No